CLINICAL TRIAL: NCT03483038
Title: A Phase II, Open-label Pilot Study Evaluating the Safety and Activity of Liposomal Irinotecan in Combination With 5-FU and Oxaliplatin in Preoperative Treatment of Pancreatic Adenocarcinoma (NEO-Nal- IRI Study)
Brief Title: A Study of the Safety and Activity of Liposomal Irinotecan in Combination With the 5-FU and Oxaliplatin in the Preoperative Treatment of Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-STO-PANC-004; IRB201800866 -A (Other: University of Florida); OCR16281 (Other: UF OnCore)
Record Dates: First submitted 2018-03-12; First posted 2018-03-29 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: pancreatic adenocarcinoma; neoadjuvant; ONIVYDE; chemotherapy; borderline resectable; resectable
MeSH Terms: interventions — irinotecan sucrosofate; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liposomal irinotecan with FOLFOX (Experimental): Subjects will receive 8 cycles and each cycle is 14 days.
  Interventions: Drug: Liposomal Irinotecan; Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Liposomal Irinotecan — Subjects will receive 60 mg/m2 intravenously on Day 1 of each 14 day cycle.
  Other Names: ONIVYDE
Drug: FOLFOX regimen — Subjects will receive FOLFOX (oxaliplatin 60 mg/m2 IV, leucovorin 400 mg/m2 IV, and 5-fluorouracil 2400 mg/m2 IV) on Day 1 of each 14 day cycle.

SUMMARY:
This is a phase II, single arm, non-randomized, open label study of liposomal irinotecan with FOLFOX in the neoadjuvant setting in patients with resectable or borderline resectable, previously untreated pancreatic adenocarcinoma. The primary objective of this study is to investigate the safety and feasibility of this treatment regimen in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age.
* A new clinical diagnosis of resectable or borderline resectable, previously untreated pancreatic adenocarcinoma confirmed by pathologic specimen evaluation
* No clinical evidence of metastatic disease
* Potentially resectable local disease, as confirmed by CT or MRI of the abdomen
* ECOG performance status of 0 or 1
* Any biliary obstruction must have been treated.
* Subjects with known or suspected Gilbert's disease must be formally tested for UGT1A1*28 with results available to study team prior to treatment initiation
* Adequate organ function; as defined by:

  i. Hematologic-
  1. ANC > 1,500 cells/μl without the use of hematopoietic growth factors; and
  2. Platelet count > 100,000 cells/μl; and
  3. Hemoglobin > 9 g/dL (blood transfusions are permitted for patients with hemoglobin levels below 9 g/dL)

     ii. Hepatic-

  <!-- -->

  1. Serum total bilirubin within 1.5 x upper limit of normal (ULN) for the institution, with a trend downwards (biliary drainage is allowed for biliary obstruction),
  2. AST and ALT less than or equal to 2.5 x ULN

     iii. Renal- Serum creatinine less than or equal to 1.5 x ULN

     iv. Cardiac- Normal ECG or ECG without any clinically significant findings as defined by the treating physician
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 7 months after the last dose of study drug to minimize the risk of pregnancy
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 4 months following the last dose of study drug.

Exclusion Criteria:

* A medical history of prior anti-cancer treatment for pancreatic cancer.
* Locally advanced unresectable disease or evidence of metastatic disease.
* Any other invasive malignancy within the past three years.
* Presence of any known contraindications to or hypersensitivities to the investigational products.
* Use of strong CYP3A4 inhibitors or inducers which cannot be discontinued prior to study entry.
* A non-surgical candidate.
* Subject is unable to understand, provide consent or comply with study requirements, treatments or instructions in the opinion of the treating physician.
* Uncontrolled diarrhea, active infection, known interstitial lung disease or other medical condition that precludes safe administration of this combination therapy consistent with manufacturer recommendations.
* Unwilling/unable to comply with birth control requirements while on study.
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 7 months for females and 4 months for males after the last dose of study drug.
* Females who are pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures.
* Known dihydrypyrimidine (DPD) deficiency

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas George, MD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - Tallahassee Memorial Health Care, Tallahassee, Florida
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singhal R, Rogers SC, Lee JH, Ramnaraign B, Sahin I, Fabregas JC, Thomas RM, Hughes SJ, Nassour I, Hitchcock K, Russell K, Kayaleh O, Turk A, Zlotecki R, DeRemer DL, George TJ. A phase II study of neoadjuvant liposomal irinotecan with 5-FU and oxaliplatin (NALIRIFOX) in pancreatic adenocarcinoma. Future Oncol. 2023 Sep;19(27):1841-1851. doi: 10.2217/fon-2023-0256. Epub 2023 Sep 27. PMID 37753702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Irinotecan With FOLFOX
Started | 45
Completed | 27
Not Completed | 18
Not completed — Subjects still in follow-up | 18

BASELINE CHARACTERISTICS:
Arm/Group | Liposomal Irinotecan With FOLFOX
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: years] | 63.133 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Had Post-operative Complications 30 Days Post-surgery
Description: To determine the percentage of subjects who had post-operative complications 30 days post-surgery. Post-operative complications considered for this outcome measure included hospital readmission, death, second surgery or interventional procedure, or major complications extending hospital stay.
Time Frame: 30 days
Population: The analyzed population for this outcome measure only include those participants who had surgery after completing study treatment with liposomal irinotecan with FOLFOX.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Liposomal Irinotecan With FOLFOX
Number analyzed (Participants) | 29
percentage of participants | 10.3 [2.2 to 27]

2. Secondary Outcome: Percentage of Subjects Who Completed All Intended Cycles of Treatment
Description: To determine the percentage of subjects that completed all eight intended cycles of treatment with liposomal irinotecan with FOLFOX.
Time Frame: 4 months
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Irinotecan With FOLFOX
Number analyzed (Participants) | 45
percentage of participants | 73.3

3. Secondary Outcome: Percentage of Subjects Who Achieved a Complete Surgical Resection (R0)
Description: To determine the percentage of subjects who achieved a complete surgical resection (R0),which is determined from review of pathology reports and inclusive of pathologic nodal status and TNM staging. A complete surgical resection (R0) has been achieved when surgical margins are microscopically negative for residual tumor.
Time Frame: 7 months
Population: The analyzed population for this outcome measure only includes those subjects who had surgery after completion of treatment with liposomal irinotecan with FOLFOX.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Liposomal Irinotecan With FOLFOX
Number analyzed (Participants) | 29
percentage of participants | 89.7 [72 to 97]

4. Secondary Outcome: Percentage of Patients Achieving a Best Overall Response of Partial or Complete Response (Objective Response Rate)
Description: To determine the percentage of patients achieving a best overall response of partial or complete response according to RECIST 1.1 criteria from the start of the treatment until disease progression/recurrence. Per RECIST 1.1 criteria, a complete response is the disappearance of all target lesions (any pathological lymph nodes [whether target or non-target] must have reduction in short axis to <10 mm). A partial response is at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters.
Time Frame: 5 months
Population: The analyzed population for this outcome measure only includes those participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Liposomal Irinotecan With FOLFOX
Number analyzed (Participants) | 38
percentage of participants | 44.7 [29 to 62]

5. Secondary Outcome: Difference Between Baseline and Maximal Nadir of Serum CA19-9 Level
Description: To determine the difference between baseline and maximal nadir of serum CA19-9 level
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units/mL
Arm/Group | Liposomal Irinotecan With FOLFOX
Number analyzed (Participants) | 45
units/mL | 756.9 (2932.7)

6. Secondary Outcome: Subject Physical, Social, Emotional, and Functional Well-being During Treatment
Description: To determine subject physical, social, emotional, and functional well-being during treatment, as measured by the FACT-G questionnaire. The FACT-G is a 27 item questionnaire where subjects respond to item with a score of 0-4. The responses to the questions are summed to calculate 4 sub-scores: physical well-being (score range 0-28), social well-being (score range: 0-28), emotional well-being (score range: 0-24), and functional well-being (score range: 0-28). The 4 sub-scores are also summed to calculate the total score. Total scores range from 0-108. A higher sub-score or total score indicates better quality of life. Participants completed the FACT-G at Cycles 1, 5, and 8, as well as at the pre-surgical evaluation and follow-up visits.
Time Frame: Cycles 1, 5, and 8 and at pre-surgical evaluation and post-surgical follow-up visits
Population: The number of participants analyzed for some sub-scores and total scores differs from the overall number of participants due to missing questionnaire responses for some participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Irinotecan With FOLFOX
Number analyzed (Participants) | 45
score on a scale
  Physical well-being (Cycle 1) | 5.1 (4.8)
  Social well-being (Cycle 1) | 24.7 (4)
  Emotional well-being (Cycle 1): number analyzed (Participants) | 44
  Emotional well-being (Cycle 1) | 8.7 (4.3)
  Functional well-being (Cycle 1): number analyzed (Participants) | 44
  Functional well-being (Cycle 1) | 19.8 (5)
  Total score (Cycle 1): number analyzed (Participants) | 44
  Total score (Cycle 1) | 58.4 (6.6)
  Physical well-being (Cycle 5): number analyzed (Participants) | 36
  Physical well-being (Cycle 5) | 8.4 (4.8)
  Social well-being (Cycle 5): number analyzed (Participants) | 36
  Social well-being (Cycle 5) | 24.2 (4.2)
  Emotional well-being (Cycle 5): number analyzed (Participants) | 36
  Emotional well-being (Cycle 5) | 7.4 (4.6)
  Functional well-being (Cycle 5): number analyzed (Participants) | 36
  Functional well-being (Cycle 5) | 18.5 (5.9)
  Total score (Cycle 5): number analyzed (Participants) | 36
  Total score (Cycle 5) | 58.5 (9.9)
  Physical well-being (Cycle 8): number analyzed (Participants) | 34
  Physical well-being (Cycle 8) | 8.1 (4.9)
  Social well-being (Cycle 8): number analyzed (Participants) | 34
  Social well-being (Cycle 8) | 24.5 (3.9)
  Emotional well-being (Cycle 8): number analyzed (Participants) | 34
  Emotional well-being (Cycle 8) | 8.3 (4.3)
  Functional well-being (Cycle 8): number analyzed (Participants) | 34
  Functional well-being (Cycle 8) | 18.3 (5.2)
  Total score (Cycle 8): number analyzed (Participants) | 34
  Total score (Cycle 8) | 59.2 (8.3)
  Physical well-being (Pre-surgical evaluation): number analyzed (Participants) | 29
  Physical well-being (Pre-surgical evaluation) | 5.9 (4.4)
  Social well-being (Pre-surgical evaluation): number analyzed (Participants) | 29
  Social well-being (Pre-surgical evaluation) | 24.5 (3.7)
  Emotional well-being (Pre-surgical evaluation): number analyzed (Participants) | 29
  Emotional well-being (Pre-surgical evaluation) | 8.1 (4)
  Functional well-being (Pre-surgical evaluation): number analyzed (Participants) | 29
  Functional well-being (Pre-surgical evaluation) | 19.1 (5.7)
  Total score (Pre-surgical evaluation): number analyzed (Participants) | 29
  Total score (Pre-surgical evaluation) | 57.6 (8.1)
  Physical well-being (Follow-up): number analyzed (Participants) | 32
  Physical well-being (Follow-up) | 8.5 (5.5)
  Social well-being (Follow-up): number analyzed (Participants) | 32
  Social well-being (Follow-up) | 24.6 (3.8)
  Emotional well-being (Follow-up): number analyzed (Participants) | 32
  Emotional well-being (Follow-up) | 7.8 (4)
  Functional well-being (Follow-up): number analyzed (Participants) | 32
  Functional well-being (Follow-up) | 15.4 (5.9)
  Total score (Follow-up): number analyzed (Participants) | 32
  Total score (Follow-up) | 56.4 (8.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until either the post-operative visit (if the subject had surgery) or until 30 days after the last dose of study treatment (if the subject did not have surgery). Adverse events were collected for up to 291 days.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator from the time of informed consent until either the post-operative visit (if the subject had surgery) or until 30 days after the last dose of study treatment (if the subject did not have surgery). Adverse events were assessed by physical examination, labs, and subject self-reports.
Arm/Group | Liposomal Irinotecan With FOLFOX
All-Cause Mortality (participants affected / at risk) | 27/45
Serious Adverse Events (participants affected / at risk) | 20/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Irinotecan With FOLFOX (N=45)
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Appendicitis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Biliary tract infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Enterocolitis infectious (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Hematoma (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 5
Neutrophil count decreased (Investigations) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Sepsis (Infections and infestations) | 1
Thromboembolic event (Vascular disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Irinotecan With FOLFOX (N=45)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 22
Agitation (Psychiatric disorders) | 2
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 4
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7
Anemia (Blood and lymphatic system disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 20
Anxiety (Psychiatric disorders) | 8
Aspartate aminotransferase increased (Investigations) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4
Biliary tract infection (Infections and infestations) | 1
Bloating (Gastrointestinal disorders) | 2
Blood bilirubin increased (Investigations) | 2
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bronchial infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Cardiac troponin I increased (Investigations) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Chills (General disorders) | 4
Constipation (Gastrointestinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 8
Depression (Psychiatric disorders) | 4
Diarrhea (Gastrointestinal disorders) | 37
Dizziness (Nervous system disorders) | 7
Dry mouth (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema face (General disorders) | 1
Edema limbs (General disorders) | 7
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Erythroderma (Skin and subcutaneous tissue disorders) | 1
Facial pain (General disorders) | 2
Fatigue (General disorders) | 36
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 5
Flatulence (Gastrointestinal disorders) | 1
Flu like symptoms (General disorders) | 1
Flushing (Vascular disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 1
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypertension (Vascular disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 22
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Infusion related reaction (General disorders) | 3
Insomnia (Psychiatric disorders) | 6
Lethargy (Nervous system disorders) | 1
Lymphocyte count decreased (Investigations) | 5
Malaise (General disorders) | 2
Mucosal infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 12
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 39
Neutrophil count decreased (Investigations) | 23
Non cardiac chest pain (General disorders) | 2
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 12
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 23
Platelet count decreased (Investigations) | 7
Presyncope (Nervous system disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Sinus tachycardia (Cardiac disorders) | 3
Sinusitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 2
Thromboembolic event (Vascular disorders) | 5
Urinary frequency (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 3
Urinary tract pain (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 17
Weight loss (Investigations) | 11
White blood cell decreased (Investigations) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT03483038/Prot_SAP_000.pdf